CLINICAL TRIAL: NCT05665530
Title: A Phase 1 Open-Label, Multi-Center, Safety and Efficacy Study of PRT2527 as Monotherapy and in Combination With Zanubrutinib or Venetoclax in Participants With Relapsed/Refractory Hematologic Malignancies
Brief Title: A Study of PRT2527 as Monotherapy and in Combination With Zanubrutinib or Venetoclax in Participants With R/R Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT2527-02
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Aggressive B-Cell Non-Hodgkin's Lymphoma (NHL); Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL); Mantle Cell Lymphoma (MCL); Richter's Syndrome; T-cell Lymphoma; Diffuse Large B-cell Lymphoma (DLBCL); Marginal Zone Lymphoma; Myeloid Malignancies; Acute Myeloid Leukemia (AML); Chronic Myelomonocytic Leukemia (CMML); Myelodysplastic Syndrome (MDS); MDS/Myeloproliferative Neoplasm (MPN) Overlap Syndrome
Keywords: Aggressive B-Cell Non-Hodgkin's Lymphoma (NHL); Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; CDK9; Cyclin-Dependent Kinase 9; Hematologic Malignancies; Mantle Cell Lymphoma (MCL); PRT2527; Relapse/Refractory; Richter's Syndrome; T-cell Lymphoma (TCL); Zanubrutinib; Diffuse Large B-cell lymphoma (DLBCL); Venetoclax; Marginal Zone Lymphoma (MZL); Myeloid Malignancies; Acute Myeloid Leukemia (AML); Chronic Myelomonocytic Leukemia (CMML); Myelodysplastic Syndrome (MDS); MDS/Myeloproliferative Neoplasm (MPN) Overlap Syndrome
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, T-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Hematologic Neoplasms; Recurrence | interventions — zanubrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PRT2527 Monotherapy in Lymphoid Malignancies (Experimental): PRT2527 will be administered by intravenous infusion once weekly at the dose level assigned during the dose escalation phase and at the defined RP2D dose for indication-specific cohorts during the dose confirmation phase.
  Interventions: Drug: PRT2527
- PRT2527/Zanubrutinib Combination in Lymphoid Malignancies (Experimental): PRT2527 will be administered by intravenous infusion once weekly at the dose level assigned during the dose escalation phase and at the defined RP2D dose for indication specific cohort during the dose confirmation phase.
  Zanubrutinib will be administered orally as combination therapy once or twice daily.
  Interventions: Drug: PRT2527; Drug: Zanubrutinib
- PRT2527 Monotherapy in Myeloid Malignancies (Experimental): PRT2527 will be administered by intravenous infusion once weekly at the dose level assigned during the dose escalation phase and at the defined RP2D dose for indication-specific cohorts during the dose confirmation phase.
  Interventions: Drug: PRT2527
- PRT2527/Venetoclax Combination in Myeloid Malignancies (Experimental): PRT2527 will be administered by intravenous infusion once weekly at the dose level assigned during the dose escalation phase and at the defined RP2D dose for indication specific cohort during the dose confirmation phase.
  Venetoclax will be administered orally as a combination therapy once daily.
  Interventions: Drug: PRT2527; Drug: Venetoclax

INTERVENTIONS:
Drug: PRT2527 — PRT2527 will be administered by intravenous infusion once weekly.
Drug: Zanubrutinib — Zanubrutinib will be provided in capsules for oral administration once or twice daily.
  Arms: PRT2527/Zanubrutinib Combination in Lymphoid Malignancies
Drug: Venetoclax — Venetoclax will be provided in tablet for oral administration once daily
  Arms: PRT2527/Venetoclax Combination in Myeloid Malignancies

SUMMARY:
This is a Phase 1 dose-escalation study of PRT2527, a potent and highly selective cyclin-dependent kinase (CDK) 9 inhibitor, in participants with select relapsed or refractory (R/R) hematologic malignancies. The purpose of this study is to evaluate the safety, tolerability, recommended phase 2 dose (PR2D), and preliminary efficacy of PRT2527 as a monotherapy and in combination with zanubrutinib or venetoclax.

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation, Phase 1 study of PRT2527, a CDK9 inhibitor, as monotherapy for participants with relapsed and refractory lymphoid and myeloid malignancies, in combination with zanubrutinib, a Bruton tyrosine kinase inhibitor (BTKi) for participants with lymphoid malignancies, or in combination with venetoclax, a B-cell lymphoma 2 inhibitor (BCL-2i) in participants with myeloid malignancies. The study will be conducted in two parts, the dose escalation phase and the dose confirmation phase for both monotherapy and combination therapy. The dose escalation phase will evaluate escalating doses of PRT2527 as a monotherapy and in combination with zanubrutinib or venetoclax until MTD is identified or when the RP2D is determined. The dose confirmation phase will evaluate indication-specific cohorts at the RP2D to confirm the dose.

Approximately 274 participants will be enrolled in the dose escalation and indication-specific, dose confirmation cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures
* Histologically or cytologically confirmed diagnosis of aggressive B-cell lymphoma subtypes, MCL, MZL, or CLL/SLL (including Richter's syndrome) based on local testing, or TCL (monotherapy only), AML, CMML, MDS, or MDS/MPN overlap syndrome that have relapsed or become refractory to or be ineligible for standard-of-care therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of < 2.
* Adequate organ function (hematology, renal, and hepatic)
* Echocardiogram (or multigated acquisition [MUGA] scan) indicating a left ventricular ejection fraction of ≥ 50%

Exclusion Criteria:

* Have active central nervous system involvement by malignancy, uncontrolled intercurrent illnesses, and active infections requiring systemic therapy
* Have undergone HSCT within the last 90 days or have graft versus host disease (GvHD) Grade > 1 at study entry
* Have severe pulmonary disease with hypoxemia
* History of another malignancy except for adequately treated non-melanoma skin cancer or lentigo maligna, superficial bladder cancer, and carcinoma in situ of the cervix without evidence of disease, and asymptomatic prostate cancer without known metastatic disease and no requirement for therapy
* Concurrent treatment or within 15 days of starting study treatment with strong CYP3A4 inhibitors
* Prior exposure to a CDK9 inhibitor
* Wait at least 5 half-lives of the agent or 14 days after their investigational or approved therapies before start of study treatment, whichever is shorter
* Mean corrected QT interval of > 470 msec following triplicate ECG measurement or history of long QT syndrome
* T-Cell leukemias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of PRT2527 | Baseline through Day 21, 28, or 35 days.
  Dose limiting toxicities will be evaluated during Cycle 1 depending on the treatment arm and intrapatient ramp-up.
Safety and tolerability of PRT2527 monotherapy and in combination with zanubrutinib or venetoclax: AEs, CTCAE Assessments | Baseline through approximately 2 years
  Safety and tolerability will be evaluated by incidence of DLTs, dose interruption, modification, and discontinuation due to adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Maximum tolerated dose (MTD)/Recommended phase 2 dose (RP2D) of PRT2527 monotherapy and in combination with zanubrutinib or venetoclax | Baseline through approximately 2 years
  The MTD/RP2D will be established for further investigation in participants with relapsed or refractory hematologic malignancies

SECONDARY OUTCOMES:
Anti-tumor activity of PRT2527 as monotherapy and in combination with zanubrutinib or venetoclax: Objective response rate (ORR) | Baseline through approximately 2 years
  Best overall response as assessed by the investigator in accordance with standard disease-specific criteria for the hematologic malignancies under study
Anti-tumor activity of PRT2527 monotherapy and in combination with zanubrutinib or venetoclax: Duration of response/Complete Response (DOR/DoCR) | Baseline through approximately 2 years
  Duration from time of first observed response to the earliest date of disease progression, as assessed by the investigator in accordance with standard disease-specific criteria for the hematologic malignancies under study, or death due to any cause, whichever occurs first
Pharmacokinetic profile of PRT2527 monotherapy and in combination with zanubrutinib or venetoclax: Maximum observed plasma concentration | Baseline through approximately 2 years
  PRT2527 pharmacokinetics will be calculated including the maximum observed plasma concentration (Cmax)
Pharmacokinetic profile of PRT2527 monotherapy and in combination with zanubrutinib or venetoclax: Area under the curve | Baseline through approximately 2 years
  PRT2527 pharmacokinetics will be calculated including the area under the plasma concentration versus time curve (AUC)
Pharmacokinetic profile of PRT2527 monotherapy and in combination with zanubrutinib or venetoclax: Time of maximum concentration | Baseline through approximately 2 years
  PRT2527 pharmacokinetics will be calculated including the time of maximum concentration (Tmax)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (5):
  - City of Hope, Duarte, California
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- Australia (4):
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria
  - Monash Health, Melbourne, Victoria
  - Linear Clinical Research Ltd, Perth, Western Australia
- Jewish General Hospital, Montreal, Quebec, Canada
- France (4):
  - Hopital Henri Mondor, Créteil
  - Claude Huriez Hospital, Lille
  - Centre Léon Bérard, Lyon
  - Institut Curie, Saint-Cloud
- Universitatsklinikum Koln, Klinik I fur lnnere Medizin, Cologne, North Rhine-Westphalia, Germany
- Italy (3):
  - lstituto Romagnolo per lo Studio dei Tumori "Dino Amadori" IRST, Meldola, FC
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant'Orsola, Bologna
  - Ospedale Santa Maria delle Croci - AUSL della Romagna, Ravenna
- Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship, Poland
- South Korea (3):
  - lnje University Busan Paik Hospital, Busan
  - Keimyung_University Dongsan Hospital, Daegu
  - Samsung Medical Center, Seoul
- Ente Ospedaliero Cantonale (EOC) lstituto Oncologico della Svizzera italiana (IOSl)- Ospedale San Giovanni (ORBV), Bellinzona, Canton Ticino, Switzerland
- The Leeds Teaching Hospitals NHS Trust, St James University Hospital, Leeds, West Yorkshire, United Kingdom